CLINICAL TRIAL: NCT02625350
Title: Glycemic Index of Instant Noodle With and Without Soup: Does Serving Method Have an Effect?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nutrifood Research Center, Jakarta, Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GI-noodle
Record Dates: First submitted 2015-12-01; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: instant noodle; water content; glycemic index; serving method

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Instant noodle without soup (Experimental): Instant noodle with 50 gram available carbohydrate per serving; cooked with 500 ml of water for 6 minutes and drained
  Interventions: Other: Instant noodle without soup
- Instant noodle with soup (Experimental): Instant noodle with 50 gram available carbohydrate per serving; cooked with 500 ml of water for 6 minutes, drained, and given additional 250 ml of water as soup
  Interventions: Other: Instant noodle with soup
- Glucose reference (Experimental): 250 ml glucose solution with 50 gram available carbohydrate per serving, used as reference
  Interventions: Other: Glucose reference

INTERVENTIONS:
Other: Instant noodle without soup — First, fasting blood glucose was measured. Then, subjects consumed the sample (instant noodle without soup) and blood sugar level were measured at 0', 15', 30', 45', 60', 90', and 120'
  Arms: Instant noodle without soup
Other: Instant noodle with soup — First, fasting blood glucose was measured. Then, subjects consumed the sample (instant noodle with soup) and blood sugar level were measured at 0', 15', 30', 45', 60', 90', and 120'
  Arms: Instant noodle with soup
Other: Glucose reference — First, fasting blood glucose was measured. Then, subjects consumed the glucose reference and blood sugar level were measured at 0', 15', 30', 45', 60', 90', and 120'
  Arms: Glucose reference

SUMMARY:
Glycemic index is commonly used as a method to determine the effect of a food to blood glucose. Despite its carbohydrate and fat content, instant noodle is very popular in Asia, including Indonesia. Based on the serving method, there are instant noodle without and with soup. Studies have shown that water content of a meal may influence glycemic response of the meal and thus have an effect on the result of GI measurement. However none specifically studied instant noodles nor the additional water content as soup (not incorporated in the food matrix). Therefore, this study aims to determine whether the serving method of instant noodle (with and without soup) may influence the glycemic response and glycemic index value of the meal.

DETAILED DESCRIPTION:
Glycemic index methods are performed according to Food and Agricultural Organization/WHO recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-40 years
* Fasting blood glucose 70-99 mg/dL
* Indonesians

Exclusion Criteria:

* Having diabetes
* Smoking
* If women, pregnant or lactating
* Being allergic to food used in this study
* Having gastrointestinal disturbance
* In regular medication
* Refusal to sign the consent form

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Changes in 2-h postprandial blood glucose level | through study completion, an average of 1 month
  blood glucose level will be measured in several time points (12-h fasting, 0 min, 15 min, 30 min, 45 min, 60 min, 90 min, and 120 min after sample consumption)

SECONDARY OUTCOMES:
Incremental area under the curve (IAUC) of postprandial blood glucose level | through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Yolanda, Ssi, Principal Investigator — Nutrifood Research Center; Lina Antono, MSc, Principal Investigator — Nutrifood Research Center; Astri Kurniati, MAppSc, Study Chair — Nutrifood Research Center

REFERENCES:
- [Background] Carbohydrates in human nutrition. Report of a Joint FAO/WHO Expert Consultation. FAO Food Nutr Pap. 1998;66:1-140. No abstract available. PMID 9743703
- [Result] Young KWH, Wolever TMS. Effect of volume and type of beverage consumed with a standard test meal on postprandial blood glucose responses. Nutrition Research 18(11): 1857-1863, 1998
- [Result] Torsdottir I, Andersson H. Effect on the postprandial glycaemic level of the addition of water to a meal ingested by healthy subjects and type 2 (non-insulin-dependent) diabetic patients. Diabetologia. 1989 Apr;32(4):231-5. doi: 10.1007/BF00285289. PMID 2759361
- [Result] Gregersen S, Rasmussen O, Winther E, Hermansen K. Water volume and consumption time: influence on the glycemic and insulinemic responses in non-insulin-dependent diabetic subjects. Am J Clin Nutr. 1990 Sep;52(3):515-8. doi: 10.1093/ajcn/52.3.515. PMID 2203255